CLINICAL TRIAL: NCT00062426
Title: A Randomized, Prospective Study Comparing Three Regimens Of Eloxatin ™ Plus Fluoropyrimidine For Evaluation Of Safety And Tolerability In First Line Treatment Of Patients With Advanced Colorectal Cancer (Tree Study)
Brief Title: Oxaliplatin and Bevacizumab (Avastin™) With Either Fluorouracil and Leucovorin or Capecitabine in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prologue Research International (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304771; PROLOGUE-SANOFI-ARD5099; SANOFI-ARD5099
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, leucovorin, and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them in different combinations may kill more tumor cells. Monoclonal antibodies, such as bevacizumab (Avastin™), can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. It is not yet known which regimen works better in treating advanced colorectal cancer.

PURPOSE: This randomized phase III trial is to see if oxaliplatin and bevacizumab work better when combined with either fluorouracil and leucovorin or capecitabine in treating patients who have metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of grade 3 and 4 toxic effects occurring within the first 12 weeks of treatment with 2 different schedules of oxaliplatin, bevacizumab (Avastin™), leucovorin calcium, and fluorouracil or with oxaliplatin, Avastin™, and capecitabine in patients with advanced colorectal cancer.
* Compare the overall response rate, progression-free survival, and time to treatment failure in patients treated with these regimens.
* Compare the composite toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive bevacizumab (Avastin™) IV over 30-90 minutes, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil (5-FU) IV over 46 hours beginning on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive Avastin™ IV over 30-90 minutes and oxaliplatin IV over 2 hours on days 1 and 15 and leucovorin calcium IV over 10 minutes and 5-FU IV over 3 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm III: Patients receive Avastin™ IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month, every 3 months for at least 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 375 patients (125 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic or recurrent disease not amenable to potentially curative treatment
* At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan

  * Histological or cytological confirmation is required for a solitary target lesion
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGPT and SGOT no greater than 3 times ULN

Renal

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 30 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No clinical evidence of congestive heart failure
* No unstable coronary artery disease

Pulmonary

* No interstitial pneumonia
* No extensive symptomatic fibrosis of the lungs

Gastrointestinal

* Able to tolerate oral medication
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No swallowing difficulties

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No other concurrent serious illness
* No uncontrolled infection
* No other concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix or any other cancer for which the patient has been off all therapy and in remission for at least 5 years
* No peripheral neuropathy
* No hypersensitivity to any of the study drugs or their ingredients
* No known dihydropyrimidine dehydrogenase deficiency
* No other medical or psychiatric disorder that would preclude giving informed consent or complying with study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic hematopoietic growth factor therapy
* No prior bevacizumab (Avastin™)

Chemotherapy

* At least 6 months since prior adjuvant fluorouracil, leucovorin calcium, and irinotecan
* No prior oxaliplatin
* No prior chemotherapy for metastatic or recurrent disease
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy unless for the control of bone pain

Surgery

* Recovered from prior surgery
* No prior organ allografts

Other

* More than 4 weeks since prior investigational drugs
* No concurrent iced mouth rinses for the prevention of stomatitis
* No concurrent cold cap alopecia prevention
* No concurrent pyridoxine
* No concurrent sorivudine or chemically-related analogues (e.g., brivudine)
* No concurrent chronic aspirin, nonsteroidal anti-inflammatory drugs, or warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Gams, MD, Study Chair — Prologue Research International; Lauri Welles, MD — Sanofi-Synthelabo
Locations (52):
- United States (52):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - California Cancer Care, Inc., Greenbrae, California
  - Valley Tumor Medical Group, Lancaster, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Hematology and Oncology Consultants, P.A., Orlando, Florida
  - Hematology Oncology Associates of theTreasure Coast - Port St. Lucie, Port Saint Lucie, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Peachtree Hematology and Oncology Consultants, P.C., Atlanta, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Cooper Cancer Institute at Cooper University Hospital, Voorhees Township, New Jersey
  - Advanced Oncology Associates, Armonk, New York
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Arena Oncology Associates, Great Neck, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - New York University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Physicians East - Quadrangle, Greenville, North Carolina
  - Raleigh Hematology/Oncology Associates, P.A. - Wake Practice, Raleigh, North Carolina
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Hematology/Oncology of Salem, Salem, Oregon
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - McCleod Cancer and Blood Center, Johnson City, Tennessee
  - Memphis Cancer Center, Memphis, Tennessee
  - West Clinic, Memphis, Tennessee
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Lone Star Oncology, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Medical Consultants, Milwaukee, Wisconsin

REFERENCES:
- [Background] Leighl NB, Bennouna J, Yi J, Moore N, Hambleton J, Hurwitz H. Bleeding events in bevacizumab-treated cancer patients who received full-dose anticoagulation and remained on study. Br J Cancer. 2011 Feb 1;104(3):413-8. doi: 10.1038/sj.bjc.6606074. Epub 2011 Jan 18. PMID 21245868